CLINICAL TRIAL: NCT01094756
Title: Central Dopamine Receptors In Obesity
Brief Title: Brain, Obesity, Dopamine and You Study
Acronym: BODY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 75-01
Record Dates: First submitted 2010-03-17; First posted 2010-03-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Psychotherapy; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese group - Group 1 (Active Comparator): If you have a BMI between 33kg - 45kg and weight under 350 lbs you could be in group 1.
  Interventions: Dietary Supplement: meal replacements, psychotherapy, dietary education
- Lean group - Group 2 (No Intervention): If you have a BMI between 18.5 kg - 24.9 kg you could be in group 2.

INTERVENTIONS:
Dietary Supplement: meal replacements, psychotherapy, dietary education — After the screening and scan days are completed, obese subjects will begin a lifestyle intervention program that includes dietary (low-calorie diet) and behavioral education topics. Treatment will be provided in individual weekly sessions. Each hour-long session will be led by a behavioral counselor or registered dietitian in the Weight Management Center at Washington University. The behavioral program will use cognitive-behavioral techniques to foster adherence to diet prescriptions and to build a supportive environment for the participant. The program will emphasize strategies of self-monitoring and goal-setting, and will include problem-solving, overcoming high-risk situations for unhealthy eating, relapse prevention, and strategies for long-term weight maintenance. Handouts will be provided for study subjects to allow them to record the setting and reaching of dietary goals, as well as summarize the key points of the educational content.
  Arms: Obese group - Group 1

SUMMARY:
Central dopamine is thought to play a significant role in obesity. In support of this idea, animal studies and one human positron emission tomography (PET) study have found reduced postsynaptic D2-like receptor availability in the striatum in obesity, with lower D2 receptor availability associated with higher weight. In addition, reward sensitivity and hedonic responses, known to be related to dopamine function, have also been implicated in obesity and obesity-related eating behavior. These reports have led to the concept that dopaminergic abnormalities (e.g. reduced D2-like receptors) influence reward sensitivity, leading to altered eating behaviors and eventually obesity. However, there are several critical limitations of the human D2 receptor studies that limit the strength of their conclusions and thus the interpretations and speculations embedded in literature that relies on this work. First, estimates of D2-like receptors in humans have been confounded by potential differences in endogenous dopamine release since the PET ligand (raclopride) used is known to be displaceable from receptors by endogenous dopamine. Second, failure to rigorously screen obese individuals for diabetes confounds conclusions, since diabetes has been independently associated with dopaminergic abnormalities such as reduced D2-like receptors and muted dopamine release in diabetic rats. Finally, no human studies have addressed whether reduced D2-like receptor levels are a risk factor for obesity, a consequence of engaging in obesity-related behaviors or being obese or all of the above.

ELIGIBILITY:
Inclusion Criteria:

* 41 obese adults (BMI 33 kg - 45 kg.)
* 24 lean adults (BMI 18.5 kg - 24.9 kg.)

Exclusion Criteria:

* Subjects who are:

  1. smokers,
  2. pregnant or lactating, postmenopausal,
  3. have diabetes or impaired oral glucose tolerance (fasting blood glucose level of < 100 mg/dl and a 2 hour post-glucose challenge plasma glucose level of < 140mg/dl, per ADA criteria; ADA 2004),
  4. significant organ system dysfunction, anemia (Hb <10 g/dl),
  5. take medications that could influence the study results, any history of dopamine agonist or antagonist treatment (e.g. neuroleptics or metoclopramide),
  6. parkinsonism on exam,
  7. borderline or lower IQ (<80 full scaled score), or
  8. any psychiatric or neurologic illness (e.g. drug abuse, Parkinson disease, Tourette syndrome, stroke) that could affect the interpretation of the data, compliance or completion of the study will be excluded. Specific psychiatric exclusions are lifetime psychosis, current mania, substance dependence, major depression, social phobia, tic disorders, eating disorders and panic disorder. Dysthymia will not be excluded, but levels of depression will be measured with the BDI for future exploratory analysis.
* Lean subjects will be excluded for being obese in the past (based on maximum BMI not related to pregnancy).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2010-07; Primary Completion 2015-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To determine the status of postsynaptic D2-like receptor binding in humans with obesity. | 1 year for each participant
  To test this hypothesis, we will measure D2-like receptor binding with PET and a specific, non-competitive D2-like receptor ligand NMB in obese and lean individuals.

SECONDARY OUTCOMES:
To determine the relationship between D2-like receptor binding, reward sensitivity and hedonic response to sweet tastes. | 1 year per participant
  To test this hypothesis we will correlate D2-like receptor binding levels in the striatum with reward questionnaires and standardized assessments of sweet taste responses within each group.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Hershey, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Medical School, St Louis, Missouri, United States